CLINICAL TRIAL: NCT00521196
Title: Phase 2 Study of the Effect of Transcranial Direct Current Stimulation (tDCS) on Pain and Headache Frequency in Migraine.
Brief Title: Migraine--Investigational Treatment of Migraine With Noninvasive Brain Stimulation. (tDCS- Migraine)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Associate Professor of Physical Medicine and Rehabilitation, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007P000145
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Migraine
Keywords: migraine; headache; chronic; pain; brain; neurology; stimulation; noninvasive; transcranial; direct; current; tDCS; tms; rTMS; BIDMC
MeSH Terms: conditions — Migraine Disorders; Headache; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline- 1 month (No Intervention): Subjects will be asked to maintain a migraine diary in which they will record the onset of each migraine, migraine-associated symptoms, migraine-associated pain, daily average pain, and daily average anxiety.
- tDCS- 1 month (Experimental): There will be 10- twenty minute sessions of the tDCS intervention over a four week period. During each tDCS session, two electrodes are placed over selected areas of the brain. 2 mA of direct current will flow through the electrodes, penetrate the scalp, and create a flow of electrical current in the brain. The subject may feel a slight itching on the scalp. The procedure will last 20 minutes. For sham tDCS, an alternate method of stimulation will be used.
  During this phase, participants will continue to maintain their migraine diary. In addition, the pain threshold of patients will be measured at the first, fifth, and tenth sessions via Thermal Sensory Analysis and Von Frey Hair tests.
  Interventions: Device: DC Stimulator (Transcranial Direct Current Stimulator)
- Follow Up- 4 months (No Intervention): During the follow up phase, subjects will meet with the study investigators a total of 5 times for follow up monitoring. Participants will continue to maintain their migraine diary during this time.
- Active tDCS- 1 month (Other): Participants randomized to sham tDCS (placebo) will be given the opportunity to receive the active intervention if the intervention is found to be safe and efficacious.
  Interventions: Device: DC Stimulator (Transcranial Direct Current Stimulator)

INTERVENTIONS:
Device: DC Stimulator (Transcranial Direct Current Stimulator) — Subjects will receive a total of 10 sessions of either active tDCS or sham tDCS over a four-week period (administered every other day during weekdays over the course of one month). During each tDCS session, two electrodes are placed over selected areas of the brain. The anode is placed on the motor cortex contralateral to the side where migraines predominant; the cathode is placed near the supraorbital area, opposite the anode. A small battery powered device drives 2 mA of direct current through the two electrodes. The direct current will flow through the electrodes, penetrate the scalp, and create a flow of electrical current in the brain. The procedure will last 20 minutes. For sham tDCS, an alternate method of stimulation will be used.
  Other Names: NeuroConn GmbH; http://www.eldith.de/products/stimulator
  Arms: Active tDCS- 1 month; tDCS- 1 month

SUMMARY:
The purpose of this study is to determine whether a painless and noninvasive procedure called Transcranial Direct Current Stimulation (tDCS) can be an effective therapy for the treatment of migraine and migraine-associated pain.

Stimulation of the motor cortex with tDCS has already been shown to relieve pain in patients with other chronic pain syndromes, including traumatic spinal cord injury and fibromyalgia. Patients with migraine are usually extremely sensitive to pain. A treatment that targets the areas of the brain that are related to the experience of pain may also help decrease pain in patients with migraine. Pain control with this localized approach may help avoid the problems due to pain medications that affect all organs in the body.

We hypothesize that 10 sessions of Transcranial Direct Current Stimulation (tDCS) applied over the area of the brain that controls pain and motor function will decrease pain and headache frequency in patients with migraine.

DETAILED DESCRIPTION:
We will rigorously test whether modulation of the motor cortex by tDCS is an effective treatment for patients with migraine through the following specific aims:

A) The primary aim of this study is to determine whether transcranial direct current stimulation applied to the motor cortex in patients with migraine induces a significant decrease in the pain associated with migraine attacks as compared with sham tDCS. We will also measure changes in the number of migraine attacks, abortive drug intake (e.g. opioids, triptans), as well as overall improvement in the quality of life to assess the effects of this treatment.

B) Determine whether the clinical effects of tDCS are long-lasting. We will therefore compare the amelioration of migraine-associated pain between active and sham tDCS after 1, 2 and 4 months of treatment.

C) Determine whether tDCS changes the threshold for pain detection as compared with sham tDCS. Patients with migraine have a lower threshold for pain as compared to healthy subjects and we hypothesize that this threshold as measured by Von Frey Hair Test and Quantitative Sensory Test will increase after stimulation with tDCS.

D) Finally, we will examine whether 1 month of tDCS treatment is safe for use in migraine patients. Safety will be assessed through neuropsychological tests and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 18 and 65 years of age.
* The diagnosis must meet the 2004 IHS criteria for migraine without aura, migraine with aura, or chronic migraine.
* The duration of the disease must be of at least one year.
* Subjects must have maintained their routine preventative medication consistently for at least two months (if applicable) prior to study initiation.

Exclusion Criteria:

* Patients with major depression with suicidal risk, as clinically defined.
* Patients with other known neuropsychiatric disorders.
* Patients with other chronic pain disorders
* History of substance abuse or dependence within the last six months
* Known brain metastasis
* History of neurological disorders (such as stroke)
* History of brain surgery
* Prior experience with tDCS
* Abnormal neurological examination, other than those pertaining to the signs of the condition studied in this protocol.
* Contraindication to tDCS: metallic hardware in the head or scalp: shrapnel, surgical clips, or fragments from welding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2012-01-13 (Actual); Study Completion 2012-01-13 (Actual)

PRIMARY OUTCOMES:
Migraine-associated pain (maximum headache intensity) | 6 months
Migraine frequency (# of headache days per month) | 6 months
Daily average pain | 6 months

SECONDARY OUTCOMES:
Thermal pain threshold | 1 month
Daily average anxiety | 6 months
Analgesic drug use | 6 months
Von Frey Hair | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, Principal Investigator — Berenson-Allen Center for Noninvasive Brain Stimulation; Beth Israel Deaconess Medical Center; Soroush Zaghi, B.S., Study Chair — Harvard Medical School; Beth Israel Deaconess Medical Center; Alexandre DaSilva, DDS, DMedSc, Study Director — Mclean Hospital
Locations (1):
- Beth Israel Deaconess Medical Center: Berenson-Allen Center for Noninvasive Brain Stimulation, Boston, Massachusetts, United States

REFERENCES:
- [Background] Fregni F, Pascual-Leone A. Technology insight: noninvasive brain stimulation in neurology-perspectives on the therapeutic potential of rTMS and tDCS. Nat Clin Pract Neurol. 2007 Jul;3(7):383-93. doi: 10.1038/ncpneuro0530. PMID 17611487
- [Background] Fregni F, Freedman S, Pascual-Leone A. Recent advances in the treatment of chronic pain with non-invasive brain stimulation techniques. Lancet Neurol. 2007 Feb;6(2):188-91. doi: 10.1016/S1474-4422(07)70032-7. PMID 17239806
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Brighina F, Piazza A, Vitello G, Aloisio A, Palermo A, Daniele O, Fierro B. rTMS of the prefrontal cortex in the treatment of chronic migraine: a pilot study. J Neurol Sci. 2004 Dec 15;227(1):67-71. doi: 10.1016/j.jns.2004.08.008. PMID 15546593
- See also: Related Info — http://tmslab.org/